CLINICAL TRIAL: NCT03873090
Title: Phase I-II Study of High Dose SBRT in 4 Fractions for Intermediate Risk Prostate Cancer
Brief Title: SBRT in 4 Fractions for Prostate Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istituto Clinico Humanitas (Other)
Responsible Party: Principal Investigator, Michele Tedeschi, Head of Clinical Trial Department, Istituto Clinico Humanitas
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1136
Record Dates: First submitted 2019-02-14; First posted 2019-03-13 (Actual); Last update posted 2019-03-13 (Actual); Status verified 2019-03

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- SBRT in 4 fraction (Experimental): Selected intermediate risk prostate cancer patients treated with 4 fraction SBRT
  Interventions: Other: SBRT

INTERVENTIONS:
Other: SBRT — hypofractionated accelerated RT for prostate cancer with FFF (Free Flattened Filter) beam. The schedule will be [ 4 x 9.5 Gy = 38 Gy ] delivered in 5 alternative days, corresponding to an NTD2 between 95 and 119 Gy for an α/β estimate between 3 and 1.5 Gy.

SUMMARY:
This is a prospective multicentric phase-I-II pilot feasibility study. The main objective is to study early and late side effects of hypofractionated accelerated RT for prostate cancer with FFF (Free Flattened Filter) beam. The schedule will be [ 4 x 9.5 Gy = 38 Gy ] delivered in 5 alternative days.

ELIGIBILITY:
Inclusion Criteria:

* Age ≤ 85years.
* WHO performance status ≤ 2.
* PSA>10 and ≤ 20 ng/ml or Gleason Score 7 or T2a-T2c.
* Histologically proven prostate adenocarcinoma
* No pathologic lymph nodes on CT/ MRI scan.
* No distant metastases.
* No previous prostate surgery other than TURP (at least 6 weeks interval before initiation of RT).
* No malignant tumours in the previous 5 years.
* IPSS 0-7.
* Combined HT according to risk factors.
* Informed consent.

Exclusion Criteria:

* Prostate size greater than 60cc.
* Previous TURP less than 6 weeks before radiotherapy.
* Previous prostate surgery other than TURP.
* Diabetes *.
* Use of anticoagulants drugs *.
* Chronic inflammatory bowel disease *.
* Previous pelvic irradiation.
* Inability to obtain written informed consent.

Ages: 18 Years to 85 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2013-06-12 (Actual); Primary Completion 2018-05-23 (Actual); Study Completion 2018-05-23 (Actual)

PRIMARY OUTCOMES:
Toxicity assessment of 4 fractions SBRT in selected intermediate risk prostate cancer patients. | up to 5 years
  Toxicity assessment: The presence and grading (CTAE v3/ EORTC-RTOG) of adverse events will be recorded.
Tumour response to local radiation therapy by assessing freedom from biochemical failure. | up to 5 years
  Tumour response is evaluated on ASTRO DEFINITION of PSA relapse (+2 from Nadir of PSA).

IPD SHARING:
Plan to Share IPD: No